CLINICAL TRIAL: NCT05724667
Title: An Evaluation of the Flippin' Pain Seminar Series: a Chronic Pain Education Campaign
Brief Title: An Evaluation of a Flippin' Pain Seminar Series
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: Connect Health Ltd (Unknown)
Responsible Party: Principal Investigator, Dr Sophie Suri, Research Associate at Teesside University, Teesside University
Other Study IDs: 2023 Jan 11120 Suri
Record Dates: First submitted 2023-01-20; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain
Keywords: Pain Science Education; Public Health; Persistent Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Flippin' Pain Seminar Series — A chronic pain education campaign

SUMMARY:
The goal of this study is to evaluate a chronic pain seminar series, Flippin' Pain. The primary aim is to examine the impact of the seminars on attendees' beliefs and perceptions of the following with regards to chronic pain: medications, surgery, physical activity, and scans. A secondary aim is to examine attendees' experience of the seminar events. Seminar attendees included people with chronic pain and on an NHS waiting list for treatment, people with chronic pain and not on an NHS waiting list for treatment, healthcare professionals and non-healthcare professionals without chronic pain.

DETAILED DESCRIPTION:
Chronic pain is defined as pain that continues for more than twelve weeks despite treatment. Chronic pain can be highly debilitating and have a devastating impact on an individual's mental and physical health and social aspects of their life. Poor understanding of chronic pain is widespread and can greatly reduce a) an individual's ability to manage their condition and b) the clinician's ability to treat the condition successfully. Educational interventions are therefore recommended. Flippin' Pain is a public health campaign that aims to improve understanding of chronic pain.

In February/March 2022, as part of the Flippin' Pain campaign, the Scottish government and NHS contracted Connect Health (TM) to deliver a series of 3 seminars in Scotland focused on pain science education. It was part of the Scottish Government 'Waiting Well' initiative and specifically targeted people on waiting lists for pain and musculoskeletal services in Scotland, although non-NHS individuals could also join including health professionals. Everyone who attended the seminars was asked if they would be happy to be contacted by the organisers as part of an evaluation of this event series.

Evaluation questionnaires were completed by 442 participants. This study will therefore be a secondary data analysis of this anonymous questionnaire data set to a). examine the impact of the seminars on attendees' beliefs and perceptions of chronic pain focusing on views towards medications, surgery, physical activity, and scans, and b). examine attendees' experience of the seminar events themselves.

The quantitative data collected from the questionnaires will be analysed using descriptive statistics. The qualitative free-text data collected from the questionnaires will be analysed using thematic analysis following Braun and Clarke's Framework.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who took part in the seminar series, answered yes to this question posed on sign-up to the seminars - 'Would you be happy to be contacted by the organisers as part of evaluation of this event series, to take part in further research into chronic pain or to provide feedback on the Flippin' Pain campaign?' and completed the evaluation questionnaire will be included in this evaluation.

Exclusion Criteria:

* Anyone who answered no to the question: 'Would you be happy to be contacted by the organisers as part of evaluation of this event series, to take part in further research into chronic pain or to provide feedback on the Flippin' Pain campaign?' provided on sign-up for the seminars will not be included in this study.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: i) People with chronic pain and on an NHS waiting list for treatment. ii) People with chronic pain and not on an NHS waiting list for treatment. iii) Healthcare professionals. iv) Non-healthcare professionals without chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Attendees' at a Flippin' Pain seminar series beliefs and perceptions of the following with regards to chronic pain - medications, surgery, physical activity, and scans. | 1-2 days post event
  Measured using a webinar evaluation questionnaire

SECONDARY OUTCOMES:
Attendees' experience of a Flippin' Pain seminar series event. | 1-2 days post event
  Measured using a webinar evaluation questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sophie V Suri, PhD, Principal Investigator — Teesside University
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymous.

REFERENCES:
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006. 3; 77-101.
- [Background] NHS Inform. [internet]. NHS. 2023 [cited 2022 Nov 6]. Available from: https://www.nhsinform.scot/illnesses-andconditions/mental-health /mental-health-self-help-guides/chronic-pain-self-help-guide
- [Background] Robinson V, King R, Ryan CG, Martin DJ. A qualitative exploration of people's experiences of pain neurophysiological education for chronic pain: The importance of relevance for the individual. Man Ther. 2016 Apr;22:56-61. doi: 10.1016/j.math.2015.10.001. Epub 2015 Oct 20. PMID 26511524